CLINICAL TRIAL: NCT02726217
Title: NYULMC-CareSmarts Study: A Pilot Study to Determine the Feasibility, Acceptability, and Potential Efficacy of an SMS-based Mobile Intervention to Enhance Type 2 Diabetes Self-management
Brief Title: NYULMC CareSmarts Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-00923
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Type 2 Diabetes (T2D)
Keywords: CareSmarts; SMS-based mobile
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CareSmarts Intervention (Experimental): Participants in the program receive text messages about diabetes self-care
  Interventions: Behavioral: CareSmarts Mobile Health Diabetes Program; Behavioral: Standard of Care Reminders and Self Assessments
- Control (Active Comparator): Standard of Care reminders and assessments for individuals with Diabetes
  Interventions: Behavioral: Standard of Care Reminders and Self Assessments

INTERVENTIONS:
Behavioral: CareSmarts Mobile Health Diabetes Program — Nurses from Diabetes Clinic will use a web-based enrollment form that includes the patient's mobile phone number, diabetes care plan, and preferred times for receiving messages. Participants in the program receive text messages about diabetes self-care. The contents of the messages that the participants receive are modified through software every two weeks as needed, based on their interactions with the system. Participants follow a flexible education curriculum in which they move from one topic to the next at their own pace.
  Arms: CareSmarts Intervention
Behavioral: Standard of Care Reminders and Self Assessments

SUMMARY:
CareSmarts is a theory-driven behavioral intervention designed to improve self-care among patients with Type 2 diabetes (T2D) with poor glycemic control (HbA1c>8%), through multiple mediators, including cuing, education, self-efficacy, social support, and health beliefs. Individuals will be randomly assigned with equal allocation to either the CareSmarts intervention or to usual care for 6 months.

DETAILED DESCRIPTION:
CareSmarts is a mobile diabetes program that provides self-management support and team-based care management for people with diabetes through automated SMS messages. The program is a theory-driven behavioral intervention designed to improve self-care through multiple mediators, including cuing, education, self-efficacy, social support, and health beliefs. Participants in the program receive educational and motivational text messages about diabetes self-care, some prompts to engage in a particular action (for example, "Time to check your blood sugar"), and some self-assessment questions (such as, "Do you need refills of any of your medications?") to which the patient responds by texting. Participants' responses to self-assessment questions are used to facilitate remote monitoring and care management by the health care team. A response that is outside established parameters triggers an alert. Using protocols, nurses respond to each alert by the next business day.

ELIGIBILITY:
Inclusion Criteria:

* have a DRG Code of T2D, and be prescribed at least one oral T2D drug and/or insulin.
* must own an SMS capable mobile device and be willing to send and receive SMS messages regarding T2D self-management.
* The participant's physician of record will have verified that his/her patient can safely participant in an intervention study that targets an HbA1c <7%.

Exclusion Criteria:

* unable or unwilling to provide informed consent
* unable to participate meaningfully in an intervention that involves use of SMS messages (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking)
* unwilling to accept randomization assignment
* pregnant, plans to become pregnant in the next 6 months, or who become pregnant during the study
* gestational diabetes
* breastfeedling
* individuals who are institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have limited control over self-management)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Measure of glucose | 3 Months
Satisfaction with Care measured by Diabetes Treatment Satisfaction Questionnaire (DTSQ). | 3 Months
Adherence to the diabetes self-management regimen using the Diabetes Self Management Questionnaire (DSMQ). | 3 Months
Acceptability of the intervention protocol will be evaluated using a satisfaction survey. | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sevick, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States